CLINICAL TRIAL: NCT00934557
Title: Multi-Centre Prospective Randomized Study on the Use of Two Different Doses of Rabbit Anti-Thymocyte Globulin for GVHD Prevention in Paediatric Patients With Haematological Malignancies Given an Unrelated Donor Haematopoietic Stem Cell Transplantation
Brief Title: Randomized Study of ATG for Graft Versus Host Disease (GVHD) Prevention in Paediatric Patients Given an Unrelated Donor Stem Cell Transplantation
Acronym: ATG FRES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Italian Association for Pediatric Hematology Oncology (Other)
Responsible Party: Professor Franco Locatelli, Foundation IRCCS Policlinico San Matteo, Pavia Italy
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: ProfGVHD1
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Paediatric Patients Affected by Haematological Malignancies and Eligible to Undergo HSCT From an Unrelated Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Good prognosis/mismatched donor/BM (Experimental)
  Interventions: Drug: ATG Fresenius
- Good prognosis/mismatched donor/PB (Experimental)
  Interventions: Drug: ATG Fresenius
- Poor prognosis/matched donor/BM (Experimental)
  Interventions: Drug: ATG Fresenius
- Poor prognosis/matched donor/PB (Experimental)
  Interventions: Drug: ATG Fresenius
- Poor prognosis/mismatched donor/BM (Experimental)
  Interventions: Drug: ATG Fresenius
- Poor prognosis/mismatched donor/PB (Experimental)
  Interventions: Drug: ATG Fresenius
- Good prognosis/matched donor/BM (Experimental)
  Interventions: Drug: ATG Fresenius
- Good prognosis/matched donor/PB (Experimental)
  Interventions: Drug: ATG Fresenius

INTERVENTIONS:
Drug: ATG Fresenius
  Arms: Good prognosis/mismatched donor/BM
Drug: ATG Fresenius
  Arms: Good prognosis/mismatched donor/PB
Drug: ATG Fresenius
  Arms: Poor prognosis/matched donor/BM
Drug: ATG Fresenius
  Arms: Poor prognosis/matched donor/PB
Drug: ATG Fresenius
  Arms: Poor prognosis/mismatched donor/BM
Drug: ATG Fresenius
  Arms: Poor prognosis/mismatched donor/PB
Drug: ATG Fresenius
  Arms: Good prognosis/matched donor/BM
Drug: ATG Fresenius
  Arms: Good prognosis/matched donor/PB

SUMMARY:
Paediatric patients affected by haematological malignancies and eligible to undergo HSCT from an unrelated volunteer will be stratified according to the degree of compatibility with their donor, the source of haematopoietic stem cells employed (BM vs. PB) and the disease phase (good vs. poor prognosis). In particular, on the basis of compatibility with their donor, patients will be allocated to 2 different arms: those transplanted from an unrelated donor either perfectly matched or with a single allelic disparity at one of the HLA loci (i.e. A, B, C, and DrB1) vs. those transplanted from an unrelated donor either with 2 allelic disparities or with an antigenic disparity at the HLA loci (i.e. A, B, C, and DrB1).

Patients enrolled in the study will be randomized to receive ATG (Fresenius) at a dosage of either 30 mg/Kg (10 mg/Kg on days -4, -3 and -2) or 15 mg/Kg (5 mg/Kg on days -4, -3 and -2).

Good prognosis patients are defined as follows: ALL in 1st CR; ALL in 2nd CR belonging to S2 group; AML in 1st CR, AML in 2nd CR and relapsed more than 6 months after stopping therapy; NHL in 2nd CR; Ph+ CML in 1st CP; refractory cytopenia.

Poor prognosis patients are defined as follows: ALL in 2nd CR belonging to the S3-S4 group; ALL in ≥ 3rd CR; AML in 2nd CR and relapsed less than 6 months after stop therapy; secondary AML; NHL in 3rd CR; Ph+ CML in 2nd CP, as well as in AP; RAEB, RAEB-t, JMML.

DETAILED DESCRIPTION:
Study rationale

Several reports have documented that patients given HSCT from an unrelated volunteer have:

* Increased incidence and severity of acute GVHD;
* Increased incidence and severity of chronic GVHD;
* Increased incidence of graft rejection;
* Increased risk of transplant-related death. The use of anti-thymocyte globulin (ATG) has been demonstrated to modulate alloreactivity of T-lymphocytes, reducing the risk of post-transplant immune complications, namely graft rejection and GVHD. However, concerns about the use of ATG exist, in particular referring to an increased incidence and severity of infectious complications, increased risk of malignancy recurrence and increased risk of EBV-related PTLD.

Design of the study Paediatric patients affected by haematological malignancies and eligible to undergo HSCT from an unrelated volunteer will be stratified according to the degree of compatibility with their donor, the source of haematopoietic stem cells employed (BM vs. PB) and the disease phase (good vs. poor prognosis). In particular, on the basis of compatibility with their donor, patients will be allocated to 2 different arms: those transplanted from an unrelated donor either perfectly matched or with a single allelic disparity at one of the HLA loci (i.e. A, B, C, and DrB1) vs. those transplanted from an unrelated donor either with 2 allelic disparities or with an antigenic disparity at the HLA loci (i.e. A, B, C, and DrB1).

Patients enrolled in the study will be randomized to receive ATG (Fresenius) at a dosage of either 30 mg/Kg (10 mg/Kg on days -4, -3 and -2) or 15 mg/Kg (5 mg/Kg on days -4, -3 and -2).

Good prognosis patients are defined as follows: ALL in 1st CR; ALL in 2nd CR belonging to S2 group; AML in 1st CR, AML in 2nd CR and relapsed more than 6 months after stopping therapy; NHL in 2nd CR; Ph+ CML in 1st CP; refractory cytopenia.

Poor prognosis patients are defined as follows: ALL in 2nd CR belonging to the S3-S4 group; ALL in ≥ 3rd CR; AML in 2nd CR and relapsed less than 6 months after stop therapy; secondary AML; NHL in 3rd CR; Ph+ CML in 2nd CP, as well as in AP; RAEB, RAEB-t, JMML.

Primary end-points

• To evaluate the influence of different ATG dosages on the incidence and severity of acute GVHD. In particular, we expect an incidence of 50% acute grade II-IV GVHD in the lower dosage (15 mg/Kg) arm, whereas we expect an incidence of 25% in the higher dosage (30 mg/Kg) arm.

Secondary end-points

* To compare the incidence of chronic GVHD in the 2 ATG dosage arms.
* To compare relapse rate in the 2 ATG dosage arms.
* To compare TRM in the 2 ATG dosage arms.
* To compare EFS in the 2 ATG dosage arms
* To compare the incidence of EBV reactivation and of EBV-related post-transplant lymphoproliferative disorders in the 2 ATG dosage arms.
* To compare the incidence of CMV reactivation in the 2 ATG dosage arms.
* To compare the incidence of adenovirus infection in the 2 ATG dosage arms.
* To compare the incidence of fungal infections in the 2 ATG dosage arms.

Study population

Patients enrolled in this study have to be affected by:

* ALL in 1st, 2nd and 3rd CR;
* AML in 1st and 2nd CR;
* NHL in 2nd and 3rd CR;
* Ph+ CML in 1st and 2nd CP, as well as in AP;
* Refractory cytopenia, RAEB, RAEB-t, JMML.

Inclusion criteria

* Unrelated donor selected using high-resolution molecular typing of HLA-A, B, C and DrB1 loci, perfectly matched or with a single allelic disparity at one of the HLA loci or with 2 allelic disparities and with an antigenic disparity at the HLA loci;
* Age comprised between 0 and 19 years;
* Life-expectancy of at least 2 months;
* Use of G-CSF mobilized PB- or BM-derived haematopoietic stem cells

Exclusion criteria

* Unrelated donor selected using high-resolution molecular typing of HLA-A, B, C and DrB1 loci, with more than one antigenic disparity or more than 2 allelic disparities at the HLA loci;
* Previous allogeneic HSCT;
* Cord blood as source of haematopoietic stem cells;
* Previous treatment with rabbit ATG in the last 3 months before HSCT;
* History of allergic reactions to rabbit ATG;
* Absence of written informed consent.

Stopping rules

* 30% mortality due to acute GVHD within the first 10 and 20 patients enrolled in the 15 mg/Kg arm;
* 80% incidence of grade II-IV acute GVHD within the first 10 and 20 patients enrolled in the 15 mg/Kg arm;
* 30% fatal infections (virus and/or fungi) within the first 10 and 20 patients enrolled in the 30 mg/Kg arm;
* 50% relapse rate within the first 10 and 20 patients enrolled in the 30 mg/Kg arm;
* 80% CMV reactivation within the first 10 and 20 patients enrolled in the 30 mg/Kg arm;
* 50% EBV reactivation within the first 10 and 20 patients enrolled in the 30 mg/Kg arm;
* 30% adenovirus reactivation within the first 10 and 20 patients enrolled in the 30 mg/Kg arm.

GVHD prophylaxis All patients will receive the combination: cyclosporine-A (Cs-A 3 mg/kg/day intravenously starting from day -2) and short-term methotrexate (MTX, 10 mg/m2 on day +1, +3, +6, and +11) for GVHD prophylaxis.

Study samples Patient randomization will be performed by the coordinating study centre in Pavia; Dr. M. Zecca will be the statistician responsible for the study. Patient enrolment was calculated by a sample size evaluation method based on the log rank test to estimate the difference in the cumulative incidence of grade II-IV acute GVHD. The minimum number of patients to be randomized was 80 per arm based on a significance level of 0.05, a study power of 0.80, and hypothesizing, for children in the lower dosage arm a grade II-IV GVHD incidence of 50% and for children in the higher dosage arm a grade II-IV GVHD incidence of 25%. Interim analysis will be performed after recruitment of the first 10, 20 and 50 patients.

Duration of the study Patients will be enrolled in approximately 24 months. Each patient must have a minimum observation time of at least 12 months. Thus, the expected study duration is 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Unrelated donor selected using high-resolution molecular typing of HLA-A, B, C and DrB1 loci, perfectly matched or with a single allelic disparity at one of the HLA loci or with 2 allelic disparities and with an antigenic disparity at the HLA loci;
* Age comprised between 0 and 19 years;
* Life-expectancy of at least 2 months;
* Use of G-CSF mobilized PB- or BM-derived haematopoietic stem cells

Exclusion Criteria:

* Unrelated donor selected using high-resolution molecular typing of HLA-A, B, C and DrB1 loci, with more than one antigenic disparity or more than 2 allelic disparities at the HLA loci;
* Previous allogeneic HSCT;
* Cord blood as source of haematopoietic stem cells;
* Previous treatment with rabbit ATG in the last 3 months before HSCT;
* History of allergic reactions to rabbit ATG;
* Absence of written informed consent.

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42
Dates: Start 2008-03

PRIMARY OUTCOMES:
incidence and severity of acute GVHD | 12 months

SECONDARY OUTCOMES:
• incidence of chronic GVHD •relapse rate •TRM •EFS •incidence of infection | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Franco Locatelli, Pavia, Pavia, Italy

REFERENCES:
- [Derived] Locatelli F, Bernardo ME, Bertaina A, Rognoni C, Comoli P, Rovelli A, Pession A, Fagioli F, Favre C, Lanino E, Giorgiani G, Merli P, Pagliara D, Prete A, Zecca M. Efficacy of two different doses of rabbit anti-T-lymphocyte globulin to prevent graft-versus-host disease in children with haematological malignancies transplanted from an unrelated donor: a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Aug;18(8):1126-1136. doi: 10.1016/S1470-2045(17)30417-5. Epub 2017 Jul 10. PMID 28705454